CLINICAL TRIAL: NCT01674413
Title: Calprotectin-Directed Humira® Maintenance Therapy, a Double-blind, Double-dummy, Randomized Controlled Trial in Crohn's Disease
Brief Title: Calprotectin-Directed Humira® Maintenance Therapy (CADHUM)
Acronym: CADHUM
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit; all patients interested simply wanted to stop medication
Sponsor: Peter Higgins (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Peter Higgins, M.D., Ph.D., MSc. Assistant Professor of Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Abbott IMM 10-0105; Abbott IMM 10-0105 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2012-08-16; First posted 2012-08-28 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Crohn's; Crohns; Inflammatory Bowel Disease; IBD; Humira; Adalimumab; Adalimumab injection; Higgins; Calprotectin; biomarkers; Gastroenterology; University of Michigan; U of M
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo/Step-Down (Placebo Comparator): 1 syringe of placebo SC q 2 weeks.
  Interventions: Drug: Placebo
- PRNLOAD Arm (Active Comparator): 160 mg/80 mg Adalimumab at Weeks 0 and 2, followed by 1 syringe SC placebo q 2 weeks (except at Weeks 12/14, 24/26, and 36/38)
  Interventions: Drug: Adalimumab PRN
- Maintenance Arm (Active Comparator): Adalimumab 40 mg q 2 weeks.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 40 mg q 2 weeks, with placebo loading of 3 syringes/1 syringe at Weeks 0/2, 12/14, 24/26, and 36/38
  Other Names: Humira
  Arms: Maintenance Arm
Drug: Adalimumab PRN — 160 mg/80 mg Adalimumab at Weeks 0 and 2, followed by 1 syringe SC placebo q 2 weeks (except at Weeks 12/14, 24/26, and 36/38), with
  * PRNLOADing of 160 mg/80 mg Adalimumab at Weeks 12/14, 24/26, or 36/38 if most recent FCP is ≥167 mcg/gram of stool,
  * Or, placebo loading of 4 syringes/2 syringes at Weeks 12/14, 24/26, and 36/38 if most recent FCP is < 167 mcg/gram of stool.
  Other Names: Humira
  Arms: PRNLOAD Arm
Drug: Placebo — 1 syringe of placebo SC q 2 weeks, with additional placebo loading of 3 syringes/1 syringe at Weeks 0/2, 12/14, 24/26, and 36/38 Weeks.
  Arms: Placebo/Step-Down

SUMMARY:
This is a study that invites adults with Crohn's disease and have been responding well to Adalimumab (Humira ®) for at least 6 months. Patients frequently discontinue maintenance medications in Crohn's disease, particularly when in remission. Patients want to know that they truly need to take a medication, yet they don't want to have flares. The purpose of this study is to see that if we monitor the patient, along with looking at changes in their stool samples, we can safely stop the maintenance medication Adalimumab for up to 48 weeks, or add as-needed dosing only, and keep them in remission.

DETAILED DESCRIPTION:
Patients frequently discontinue maintenance medications in Crohn's disease, particularly when in remission. Patients want to know that they truly need to take a medication, yet they don't want to have flares. As a biomarker, fecal calprotectin < 167 has a 100% negative predictive value for flare within the next 12 weeks (Gisbert, 2009). Adalimumab has low antigenicity, and can be safely stopped and restarted later with good clinical effect (Colombel, 2007). Patients want intermittent therapy, if it can be delivered in a timely fashion when pre-clinical inflammation starts, in order to avoid clinically-significant flares. This study will combine monitoring for pre-clinical inflammation with fecal calprotectin and as-needed dosing with Adalimumab to maintain remission in patients who have obtained remission with Adalimumab. This will be compared to two comparator arms: standard maintenance therapy and complete cessation of therapy (Step-Down approach).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years of age or older at the time of informed consent.
2. Crohn's disease confirmed by endoscopy with biopsies.
3. On maintenance Adalimumab at a dose of 40 mg SC q 2 weeks without concomitant immunosuppressive therapy.
4. Must be in clinical remission (CDAI <150) at the baseline/randomization (Week 0) visit and biologic remission (both CRP <0.8 and FCP <167)at Week 0.
5. Prior medication for Crohn's disease may include one of the following and must have been stopped with wash out periods: Methotrexate, Azathioprine, 6-Mercaptopurine, Tacrolimus, Steroids.
6. Negative for TB, Hepatitis B-negative, and negative stool for Clostridium difficile.

Exclusion Criteria

1. Unable to consent for themselves.
2. Are prisoners, students or employees of the investigators, or mentally incapacitated.
3. Are unwilling to complete this 48 week study, provide stool samples throughout, or unwilling to undergo multiple venipunctures.
4. Have a current infection with Clostridium difficile, clinically-significant intestinal stricture, history of allergy, or adverse reaction, to Adalimumab, history of sensitivity to latex.
5. Are currently using steroids or systemic immunomodulators (MTX, AZA, 6-MP, or Tacrolimus), or have used another biologic medication in the past 12 weeks other than Adalimumab, or have current or past use of Kineret® (Anakinra) or Tysabri® (natalizumab).
6. Have received any live bacterial or viral vaccinations ≤ 12 weeks prior to Week 0 and must not receive 12 months after study as well as BCG vaccination
7. Are known to have congestive heart failure.
8. Have a history of, or ongoing chronic or recurrent infectious disease, including but not limited to chronic renal, chest infection (i.e. bronchiectasis) or urinary tract infection (i.e. recurrent pyelonephritis) or open, draining, or infected skin wounds or ulcers.
9. Have evidence of current clinically active and important infection.
10. Have or ever had a non-tuberculous mycobacterium infection or serious opportunistic infection (i.e. cytomegalovirus, Pneumocystis carinii, aspergillosis).
11. Are known to be infected with HIV, Hepatitis B, or Hepatitis C.
12. Have severe, progressive, or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof.
13. Have a known history of lymphoproliferative disease including lymphoma. Have a history of certain malignancies within five years of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percent Time in Remission (PTIR) in PRNLOAD vs. Placebo arms | 48 weeks
  Determine whether adding as-needed q 12 weeks Adalimumab re-loading (160 mg/80 mg) when FCP ≥167 mcg/gram of stool can improve the maintenance of remission in Crohn's disease patients who stop Adalimumab therapy (PRNLOAD Arm) compared to the placebo arm. Endpoint: Percent time in remission (q 4 week evaluation for 48 weeks).

SECONDARY OUTCOMES:
Percent Time in Remission MAINT vs. PRNLOAD | 48 weeks
  Compare the percent of monitoring visits in which the subject is in remission in each arm between the MAINT and PRNLOAD arms.
Percent Time in Remission MAINT vs. PBO | 48 weeks.
  Compare the percent of monitoring visits in which the subject is in remission in each arm between the MAINT and PBO arms.
Strict Biologic Remission Rates | 48 weeks
  Percent of visits with strict biologic remission (FCP <50 and CRP <0.5) with 3 comparisons: PRNLOAD vs. PBO, MAINT vs. PRNLOAD, MAINT vs. PBO
Subject acceptability | 48 weeks
  Measure subject acceptability of repeated stool sampling.
Subject preference | 48 weeks
  Measure subject preference for the MAINT versus PRNLOAD regimen.
Equivalence of Percent Time in Remission | 48 weeks
  Compare percent time in remission (CDAI <150) over 48 weeks, evaluation every 4 weeks across 3 arms (chi square test).
Comparison of Average CDAI | 48 weeks
  Compare average CDAI over 48 weeks, evaluation every 4 weeks across 3 arms (ANOVA).
Comparison of average IBDQ | 48 weeks
  Compare average IBDQ over 48 weeks, evaluation every 4 weeks across 3 arms (ANOVA).
Comparison of average FCP | 48 weeks
  Compare average FCP over 48 weeks, evaluation every 12 weeks across 3 arms (ANOVA).
Comparison of average CRP | 48 weeks
  Compare average CRP over 48 weeks, evaluation every 12 weeks across 3 arms (ANOVA).
Comparison of Rates of Hospitalization | 48 Weeks
  Comparison of Rates of Hospitalization across all 3 arms - hospital admissions per patient over 48 weeks (ANOVA).
Comparison of Rates of Emergency Department visits | 48 Weeks
  Comparison of Rates of Emergency Department visits across all 3 arms - hospital admissions per patient over 48 weeks (ANOVA).
Comparison of Rates of Physician visits | 48 Weeks
  Comparison of Rates of Physician visits across all 3 arms - hospital admissions per patient over 48 weeks (ANOVA).
Comparison of mg prednisone prescribed | 48 Weeks
  Comparison of average milligrams of prednisone prescribed across all 3 arms - over 48 weeks (ANOVA).

OTHER OUTCOMES:
Anti-Adalimumab antibodies | 0, 48 weeks
  Measure anti-Adalimumab antibody titers in patients at week 0 and 48 weeks (or exit visit). Compare average titers across 3 arms (ANOVA)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Higgins, MD, PhD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
no data collected